CLINICAL TRIAL: NCT03056976
Title: Cost-effectiveness of Implant Treatment for the Edentulous Mandible
Acronym: CEAIMPLANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Associate Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFG_SAP_41429
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Edentulous Mouth
Keywords: Overdenture; Dental implant; Complete denture; Cost analysis
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness of thre competing strategies for the edentulous mandible using implants
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single-implant mandibular overdenture (Experimental): A single midline implant and an O'ring/ball attachment to retain a mandibular overdenture
  Interventions: Device: Single-implant mandibular overdenture
- Two-implant mandibular overdenture (Experimental): Two implants in the canine region and two O'ring/ball attachments to retain a mandibular overdenture
  Interventions: Device: Two-implant mandibular overdenture
- Fixed mandibular denture (Experimental): A fixed four-implant mandibular denture
  Interventions: Device: Fixed mandibular denture

INTERVENTIONS:
Device: Single-implant mandibular overdenture — Complete mandibular denture retained by a single midline implant
  Other Names: Single-implant overdenture
  Arms: Single-implant mandibular overdenture
Device: Two-implant mandibular overdenture — Complete mandibular denture retained by two implants in the canine region
  Other Names: 2-implant overdenture
  Arms: Two-implant mandibular overdenture
Device: Fixed mandibular denture — A fixed mandibular denture retained by four implants
  Other Names: Full-arch mandibular prothesis
  Arms: Fixed mandibular denture

SUMMARY:
The aim of this study is to assess the cost-effectiveness of the mandibular overdenture retained by one and two implants and the mandibular fixed prosthesis retained by four implants, based on a randomized clinical trial.

DETAILED DESCRIPTION:
This randomized clinical trial alongside a cost-effectiveness analysis will include 48 edentulous individuals who meet eligibility criteria. Participants will receive conventional complete denture treatment and will be randomized into three groups: single-implant mandibular overdenture group, mandibular overdenture retained by two implants, and fixed mandibular prosthodontics retained by four implants. CBCT and panoramic radiographs will be obtained to assess if bone sites in three-dimensional terms have a minimum volume for receiving implants of at least 3.75 x 9 mm. All patients will receive Titamax IT Cortical implants (Neodent, Curitiba, Brasil) and correspondent prosthodontic components - O'ring/ball abutments for overdentures. Satisfaction with the dentures and oral health-related quality of life impacts will be considered the measures of effectiveness for the three interventions. Cost assessment and cost-effectiveness analysis will be performed from the healthcare provider perspective. Further analysis will be performed using the patient's perspective, in which the costs will be estimated according to the reference price of dental procedures and treatments of the Brazilian Dental Association (Hierarchical Brazilian Classification of Dental Procedures - CBHPO) and the gross costs will be obtained from a panel of experts. Quantification and costing of the resources will be carried out in three steps: identification of the relevant costs to the assessment; measurement of the resources used; and valuation of the resources. The costs will be calculated in Brazilian currency for each patient until one year after treatment. Incremental cost-effectiveness ratios will be calculated to assess the incremental cost for each unit of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications for implant surgery (mainly related to uncontrolled systemic diseases)
* Present enough bone volume in the mandible for implant placement without the need of bone augmentation procedures.
* Be able to understand and answer the questionnaires used in the study
* Agree to participate by providing a written informed consent.

Exclusion Criteria:

* Noncompliant participants
* Individuals who do not agree to be randomly allocated to the treatment study group
* Presence of signs of untreated temporomandibular disorders, uncontrolled systemic or oral conditions that require additional treatments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the dentures | 1-year
  A 10 cm uninterrupted visual analogue scale will be used in order to assess the participants' ratings of their satisfaction with the upper and lower dentures in relation to the parameters "general satisfaction", "comfort", "stability", "aesthetics", "ability to speak" and "ability to chew".
Oral health-related quality of life impacts | 1-year
  Oral Health Impact Profile Instrument for edentulous subjects (OHIP-EDENT) in order to assess the impact of oral health conditions on quality of life of participants.

SECONDARY OUTCOMES:
Masticatory efficiency | 1-year
  Masticatory efficiency will be assessed as a secondary outcome using a two-colored chewing gum test and a qualitative and quantitative colourimetric method to measure the color-mixing ability.
Cost | 1-year
  Direct and indirect treatment costs

CONTACTS AND LOCATIONS:
Overall Officials: Enilza Paiva, PhD, Study Chair — Dean of the Dental School, Federal University of Goias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nogueira TE, Esfandiari S, Leles CR. Cost-effectiveness analysis of the single-implant mandibular overdenture versus conventional complete denture: study protocol for a randomized controlled trial. Trials. 2016 Nov 4;17(1):533. doi: 10.1186/s13063-016-1646-0. PMID 27814749